CLINICAL TRIAL: NCT03518905
Title: Radiofrequency Ablation for the Treatment of Large Symptomatic Heterotopic Gastric Mucosa - a Prospective Randomized Sham-controlled Trial - the RAGE Study
Brief Title: Radiofrequency Ablation for the Treatment of Large Symptomatic Heterotopic Gastric Mucosa
Acronym: RAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Ivan Kristo, MD, Attending surgeon, Vize-Chair of the esophageal functional testing laboratory, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1340/2017
Record Dates: First submitted 2018-04-15; First posted 2018-05-08 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Esophagus Disorder
MeSH Terms: conditions — Esophageal Diseases | interventions — Radiofrequency Ablation; Esophagoscopy

STUDY DESIGN:
Intervention Model Description: randomized sham-controlled
Who Masked: Participant
Masking Description: Patients are blinded either to sham or treatment and unblinded after 24 weeks after final examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham-treatment (Sham Comparator): Patients with symptomatic large heterotopic gastric mucosa receive an esophagoscopy without radiofrequency ablation under sedation
  Interventions: Procedure: esophagoscopy
- treatment arm (Active Comparator): Patients with symptomatic large hetertotopic gastric mucosa receive an esophagoscopy with radiofrequency ablation (12J/cm2) using the Barrx channel RFA endoscopic catheter (Medtronic)
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — Radiofrequency ablation is performed using the Barrx Channel endoscopic catheter (Medtronic, Dublin, Republic of Ireland) generating an energy density level of 12 Joule/cm2. The energy is applied using a simplified protocol of three ablations without removal of coagulated tissue. The device is used on a routinely basis all around the world and already approved. The ablation catheter is applied through the working channel of the endoscope.
  Arms: treatment arm
Procedure: esophagoscopy — Patients receive an esophagoscopy without radiofrequency ablation under sedation
  Arms: sham-treatment

SUMMARY:
The heterotopic gastric mucosa found in the cervical esophagus was first described in 1805 and affects 10-15% of individuals undergoing esophagogastroduodenoscopy. It leads to laryngopharyngeal reflux (LPR), which causes symptoms like globus sensation, hoarseness and chronic cough. The Reflux Symptom Index (RSI) that ranges from 0-45 measures LPR. Scores greater than 13 are considered to be pathologic. Currently, patients that suffer from symptoms of LPR and present with a heterotopic gastric mucosa are routinely offered radiofrequency ablation (RFA) as curative treatment. Up to now, around 40 patients were already treated at the department of Surgery with 90% histologic eradication rates after 2 treatment sessions and no reported serious adverse event. Nevertheless, the placebo effect could also be responsible for perception of improving symptoms. Therefore, this prospective sham-controlled trial was designed to exclude the placebo effect. As the device is already approved and routinely used for focal ablation safety data are already available. Up to now, there were no major adverse events, whereas only 10% of patients describe a sensation of irritated throat that dissolves within the first three days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven presence of heterotopic gastric mucosa,
* pathologic Reflux Symptom Index (>25)
* age: 18-70
* presence of symptoms > 6 months,
* no effect on the Reflux Symptom Index to 12 weeks of standard dose proton pump inhibitor treatment
* negative symptom correlation for symptoms with reflux events in ambulatory pH monitoring

Exclusion Criteria:

* Not willing to participate in this study
* pregnancy
* lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-09-16 (Estimated); Study Completion 2020-12-16 (Estimated)

PRIMARY OUTCOMES:
Normalization of the Reflux Symptom Index | 6 months after first RFA treatment/or sham procedure
  Normalization of the Reflux Symptom Index (RSI <14) after two treatment/sham sessions evaluated 3 months after the second (sham-) treatment (therefore 6 months after the first endoscopy with/without RFA). Proton-pump inhibitors are paused 8 weeks before assessment

SECONDARY OUTCOMES:
Histological eradication rate after radiofrequency ablation or sham treatment | 6 months after first RFA treatment/or sham procedure
  Histologic eradication rate after RFA treatment/sham procedure measured after finalization of RFA (normalization of Reflux Symptom Index/or a maximum of two treatment sessions) or at the time of second sham treatment.
SF-12 quality of life | At enrollment (therefore before ablations or sham treatment) and 6 months after first radiofrequency ablation/sham treatment
Reflux Finding Score | Evaluated at the first intervention at study completion after 6 months
  the Reflux Finding Score is measured by using laryngofibroscopy to document potential absence of laryngopharyngeal reflux. The reflux finding score (RFS) represents an objective and validated instrument to analyze physical findings and severity of laryngopharyngeal reflux. An 8-item checklist with excellent inter-observer reliability grades abnormalities documented during laryngoscopy from 0-26 points. The total score is reported and summed from an 8 item checklist providing 0-4 points. Statistically, total scores greater than 7 have a likelihood of 95% to reflect LPR. Higher scores represent worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No